CLINICAL TRIAL: NCT05662384
Title: A Multicenter Prospective Study on Small Bowel Obstruction
Brief Title: Small Bowel Obstruction. A Prospective Multicener Study
Acronym: SBO
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Collaborators: North Estonian Medical Center (Unknown)
Responsible Party: Principal Investigator, Liis Jaanimäe, General Surgeon, PhD student, University of Tartu
Other Study IDs: 21010
Record Dates: First submitted 2022-12-04; First posted 2022-12-22 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Small Bowel Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized with small bowel obstruction: Patients hospitalized with a certain diagnosis during a certain period of time
  Interventions: Other: No intervention is planned

INTERVENTIONS:
Other: No intervention is planned — Observational study, no intervention

SUMMARY:
To get an overview of patients hospitalized with mechanical small bowel obstruction and the evaluate the use of contrast media as part of conservative management. To analyze how many patients were operated on and in how many cases conservative measures helped.

DETAILED DESCRIPTION:
This is a multicenter prospective study conducted at two regional hospitals of Estonia: Tartu University Hospital and North Estonian Medical Center. The data of the patients' hospitalized for SBO between May 2021 and April 2022 were collectedafter patients gave their informed consent to be enrolled in the study.

Eligible patients were adults aged 18 years or older with mechanical small bowel obstruction. Patients younger than 18 years, patients with large bowel obstruction or dynamic small bowel obstruction and/or patients who had undergone abdominal/pelvic surgery within 4 weeks of admission were excluded from the study.

Characteristics of abdominal pain (absent/intermittent/permanent), presence of nausea/vomiting, absence of flatus, results of blood tests (white blood cell count (WBC), C-reactive protein (CRP), lactate level (Lac), estimated glomerular filtration rate (eGFR)), radiology imaging techniques used, previous abdominal/pelvic surgeries, previous episodes of bowel obstruction. It was documented whether immediate surgical treatment was implemented, or whether conservative management was initiated. In the case of conservative treatment, it was recorded whether contrast media (CM) was or was not used. In the case of surgical treatment, the type of surgery (adhesiolysis/ bowel resection/ other) was recorded.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older with mechanical small bowel obstruction who signed an informed consent form

Exclusion Criteria:

* Patients younger than 18 years, patients with large bowel obstruction or dynamic small bowel obstruction and/or patients who had undergone abdominal/pelvic surgery within 4 weeks of admission were excluded from the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with mechanical small bowel obstruction
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Resolution on SBO | Hospitalization period (approximately 5 days)
  Resolution of small bowel obstruction (passing gas/flatus, contrast media in the colon on the X-ray )

CONTACTS AND LOCATIONS:
Overall Officials: Liis Jaanimäe, Principal Investigator — University of Tartu
Locations (1):
- Tartu University Hospital, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: Undecided
Patients identification numbers will be pseudonymed- the key is in a secure server and will only be accessed through smart-ID identification